CLINICAL TRIAL: NCT04529434
Title: Star Homes - Better Health Through Better Housing: Phase 2 House Evaluation
Brief Title: Star Homes Project 2
Acronym: SHP2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); CSK Research Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MAL19012
Record Dates: First submitted 2020-08-06; First posted 2020-08-27 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Malaria; Respiratory Tract Infection Acute; Diarrhoea;Acute
Keywords: Healthy houses; Tanzania
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: This is an open-label household randomised controlled trial that will compare the 110 novel-design houses with 440 traditional African homes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Households living in novel-design houses.
  Interventions: Other: Star Homes
- Arm 2 (Other): Households living in traditional African houses.
  Interventions: Other: Traditional African houses

INTERVENTIONS:
Other: Star Homes — 110 identical novel-designed houses, known as Star Homes, include the critical structural components e.g. building orientated to provide optimal shading throughout the day, light-weight & durable roof, facade and openings screened from insects to reduce insect entry while assuring airflow, an outdoor fly-proof latrine, and solar power providing electric light at night etc.
  Arms: Arm 1
Other: Traditional African houses — A traditional mud house: with wattle and daub walls, a thatched roof, and no electricity or piped water supply.
  Arms: Arm 2

SUMMARY:
Malaria, pneumonia and diarrhoea causes a lot of illness in children in Tanzania and the study want to find better ways of protecting people against these diseases and want to find out if the type of house design can affect the general health of children living in the house.

DETAILED DESCRIPTION:
The study hypothesis is that healthy houses will reduce the incidence of malaria, respiratory diseases and diarrhoeal diseases in children compared with traditional houses. And healthy houses are also likely to reduce the incidence of all-cause morbidity incidence, disease severity, improve growth and well-being. The primary endpoints will be assessed in children under 13 years of age through weekly household visits for three years. All homes will have access to basic vector control, such as insecticide treated nets (ITNs). Access to early diagnosis and appropriate malaria treatment will be assured. Approximately 2,750 Tanzanians living in 550 houses in Mtwara region, of which 110 are new design houses (Star Homes) and the remaining 440 traditional African houses will be participating in this study. 330 children living in the novel design houses and 1320 children in traditional homes will be followed for three years for the assessment of malaria, respiratory tract infections and diarrhoea. Mosquito density will be assessed from all 550 houses where tent/light trap will be used for mosquito catch at night in all study houses. Acceptance of the novel designed houses will be assessed using mixed methods. Acceptability surveys will be conducted with 550 household heads concurrently with in-depth interviews with 30 purposively selected heads of the households in the intervention arm. Ten focus group discussions will be conducted each comprising 10 heads of households making it to be 100 heads of households.

Funder: Hanako Foundation, Singapore

ELIGIBILITY:
Inclusion Criteria

Main study

* Children, aged under 13 years old, male or female
* Residing in a study village for at least 3 years
* Parents/guardian is willing and able to give written informed consent for the child to participate in the baseline and end-of study evaluation and the surveillance for malaria, respiratory tract infection and diarrhoeal disease.
* Additionally, children 10, 11, and 12 years of age provide assent to participate.

Ancillary studies

* Head of a household or other family member of a household that is taking part in the main study
* 18 years and above
* Consent to take part in the main study
* Residing and live in the village for 3 years or more
* Live in the intervention or comparison houses or a trusted community member (community leaders, medical officer and community health worker)

Exclusion criteria

Main study

* Any participant who refuses, or in the case of children whose parents/guardian refuses, to participate in the study.
* Any child who is between 10 and 12 years who refuses to provide assent
* If the family plans for moving to other village during the study period
* Parents/guardians have mental health problems

Ancillary studies

* Under 18 years
* Not provide consent
* Not living in the study village for 3 years or more

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2750 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of malaria in children under 13 years of age. | Approximately 3 years
  The incidence per year of malaria in children under 13 years old.
Incidence of respiratory tract disease in children under 13 years of age. | Approximately 3 years
  The incidence per year of respiratory tract disease in children under 13 years old.
Incidence of diarrhoeal disease in children under 13 years of age. | Approximately 3 years
  The incidence per year of diarrhoeal disease in children under 13 years old.

SECONDARY OUTCOMES:
Mean number of female An. gambiae s.l. | Approximately 3 years
  Mean number of female An. gambiae s.l./light trap/night
Mean number of flies | Approximately 3 years
  Mean number of flies/sticky trap/week in kitchens of the houses
Entomological inoculation rate of malaria vectors. | Approximately 3 years
  Compare entomological inoculation rate of mosquito inside novel and traditional rural houses.
Children requiring hospital admission | Approximately 3 years
  Compare hospitalization rate of children under 13 years living inside novel and traditional rural houses.
Major respiratory pathogens | Approximately 3 years
  From children requiring hospital admission, the most frequently detected respiratory tract pathogens will be assessed through blood culture.
Major enteric pathogens | Approximately 3 years
  From children requiring hospital admission, the most frequently detected enteric pathogens will be assessed through rotavirus ELISA testing and bacterial culture of stool specimens.
Prevalence of malaria parasitaemia among children living in novel design houses and traditional homes. | Approximately 3 years
  Prevalence will be assessed from a cross-sectional surveys of children, based on dried blood smears will be collected for quantitative polymerase chain reaction once per quarter.
Mean changes in weight | Approximately 3 years
  Weight in kilograms of children under 13 years of age recorded at baseline, annually and at end of the study.
Mean changes in height | Approximately 3 years
  Height in meters of children under 13 years of age recorded at baseline, annually and at end of the study.
Mean changes in body mass index (BMI) | Approximately 3 years
  BMI in Kg/m2 in meters of children under 13 years of age recorded at baseline, annually and at end of the study.
Mean changes in mid-upper arm circumference | Approximately 3 years
  Mid-upper arm circumference in millimeters of children under 13 years of age recorded at baseline, annually and at end of the study.
Disease severity | Approximately 3 years
  A subgroup analysis of children requiring hospital consultation and children requiring hospitalization.
Indoor temperature | Approximately 2 years
  Temperature will be measured using data loggers.
Humidity | Approximately 2 years
  Humidity will be measured using data loggers.
Carbon dioxide (CO2) | Approximately 2 years
  Carbon dioxide (CO2) will be measured using data loggers.
Particulate matter 2.5 (PM2.5) particle pollution | Approximately 2 years
  PM2.5 particle pollution will be measured using data loggers.
Acceptability of the novel design houses. | Interviews at 6 months after moving in, 1 year and at the end of the study
  The acceptability will be measured through a mixed method: 1) quantitative method i.e. closed ended questions with a pre-determined set of choices 2) qualitative method i.e. open ended questions through focused group discussions and in-depth interviews.
Bednet use | Annually (for three years)
  Assessed by asking residents and in children with less than 5 years old in traditional and novel design homes regarding the use of insecticide treated bednets.
Life-cycle analysis | Over 36 months period starting from moving in date.
  This is the cost of illness averted by living in a novel-designed home against a background of complete coverage with insecticide-treated nets. The analysis will include cost comparison (construction and maintenance of novel and control houses) and market analysis.
Durability | End of year 1, 2 and 3.
  Yearly inspections of houses (control and intervention). Maintenance of structural problems on demand.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz von Seidlein, Ass.Prof., Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- CSK Research Solutions, Dar Es Salaam, Mtwara, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be under the custodianship of MORU. With participant's consent, data from this study may be shared in a de-identified form with other groups or researchers in accordance with the MORU Data Sharing Policy.
Time Frame: After completion of trial activities and reporting
Access Criteria: MORU Data Sharing Policy. (http://www.tropmedres.ac/data-sharing-policy)

REFERENCES:
- [Derived] Mmbando AS, Ngonzi AJ, Mshamu S, Bradley J, Bojstrup TC, Ngowo HS, Knudsen J, von Seidlein L, Okumu FO, Lindsay SW. Effect of a novel house design (star home) on indoor malaria mosquito abundance in rural Tanzania: secondary outcomes of an open-label, household, randomised controlled trial. Lancet Planet Health. 2025 Apr;9(4):e253-e263. doi: 10.1016/S2542-5196(25)00046-4. PMID 40252672
- [Derived] Mshamu S, Mmbando A, Meta J, Bradley J, Bojstrup TC, Day NPJ, Mukaka M, Okumu F, Olotu A, Pell C, Deen J, Knudsen J, Lindsay SW, von Seidlein L. Assessing the impact of a novel house design on the incidence of malaria in children in rural Africa: study protocol for a household-cluster randomized controlled superiority trial. Trials. 2022 Jun 20;23(1):519. doi: 10.1186/s13063-022-06461-z. PMID 35725486